CLINICAL TRIAL: NCT06092398
Title: Role of Autologous Platelet Rich Plasma(PRP) Injection and Platelet Rich Fibrin Glue(PRFG) Interposition for Treatment of Anal Fistula
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hassan Thabet Ahmed, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRP and PRFG in anal fistula
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP and PRFG in anal fistula (Experimental): the tract fistula was cleaned with betadine 10% before PRP and PRFP were applied. Then, 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. The operation time was about 20-30 minutes, the clot formation usually takes about 8 minutes, but the anesthesia was extended to 20 minutes to make sure a complete clot in the place
  Interventions: Other: PRP and PRFG in treatment of anal fistula

INTERVENTIONS:
Other: PRP and PRFG in treatment of anal fistula — The tract fistula was cleaned with betadine 10% before PRP and PRFP were applied. Then, 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. The operation time was about 20-30 minutes, the clot formation usually takes about 8 minutes, but the anesthesia was extended to 20 minutes to make sure a complete clot in the place of fistula

SUMMARY:
To evaluate the autologous platelet rich plasma and platelet rich fibrin glue effect on the treatment of anal fistula

To asses role of platelet rich plasma and platelet rich fibrin glue in decreasing recurrence of perianal fistula

DETAILED DESCRIPTION:
An anal fistula (AF) is a tunnel connecting the anal canal or rectum (internal opening) with the skin (external opening) around the anus. Patients who have a perianal abscess have symptoms include discomfort, trouble sitting, and pus or blood discharge. Simple and complicated anal fistulas are the two types that exist. A complex fistula is difficult to manage, has a higher risk of recurrence rates, and poses a greater threat to continence after surgery. AF was associated with significant morbidity which is a devastating condition with profound effects on both the physical and psychological health of the patient.

Fibrin glue (also called fibrin sealant) is a surgical formulation used to create a fibrin clot for hemostasis, cartilage repair surgeries or wound healing. It contains separately packaged human fibrinogen and human thrombin. New procedures were published in the scientific literature, each with advantages and disadvantages. According to reports, an effective therapy option is the autologous fibrin glue that is rich in platelets.

PRP began to be used in surgery as a regenerative tissue factor

The tract fistula was cleaned with betadine 10% before PRP and PRFP were applied. Then, 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. 2 ml of PRP was injected around the fistula into the tissue (the penetration depth in injection was 5-6 mm), and 4 ml PRFP was mixed with 1 m thrombin and interpositioned into the tract. The operation time was about 20-30 minutes, the clot formation usually takes about 8 minutes, but the anesthesia was extended to 20 minutes to make sure a complete clot in the place of fistula

ELIGIBILITY:
Inclusion Criteria:

* 60 patients with perianal fistula were in the age group between 20 to 60 years old

Exclusion Criteria:

* Thrombocytopenia
* Patient with rectovaginal fistula
* fistula with chronic cavities
* Acute sepsis and patient were not willing undergo this type of treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
evaluate effect of autologous platelet rich plasma and platelet rich fibrin glue in decreasing recurrence rate of anal fistula | 3 year
  evaluate effect of autologous platelet rich plasma and platelet rich fibrin glue in decreasing recurrence rate of anal fistula

SECONDARY OUTCOMES:
to evaluate the role of platelet rich plasma and platelet rich fibrin glue in decreasing post operative complication of anal fistula | 3 year
  to evaluate the role of platelet rich plasma and platelet rich fibrin glue in decreasing post operative complication of anal fistula

CONTACTS AND LOCATIONS:
Overall Officials: maha atwa, PHD, Study Chair — Assiut University

REFERENCES:
- [Background] Abdollahi, Abbas, Elaheh Emadi, and Dariyoush Hamidi Alamdary.
- [Background] Yeung JM, Simpson JA, Tang SW, Armitage NC, Maxwell-Armstrong C. Fibrin glue for the treatment of fistulae in ano--a method worth sticking to? Colorectal Dis. 2010 Apr;12(4):363-6. doi: 10.1111/j.1463-1318.2009.01801.x. Epub 2009 Feb 7. PMID 19220380
- [Result] Ji, Lijiang, et al.